CLINICAL TRIAL: NCT01050049
Title: The Effect of Implementing Hyper-acute Stroke Guidelines on Decision-Making for or Against Thrombolytic Therapy for Stroke in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Temple University (Other)
Responsible Party: Nina T. Gentile, MD, Temple University
Other Study IDs: 11959
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2008-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Before guidelines implemented
- After guidelines implemented

SUMMARY:
The objective of this study is to determine if the implementation of guidelines utilizing immediate CT Perfusion and CT Angiography in addition to non-contrast CT alters (reduces or increases) the time to decision-making for or against rt-PA in acute ischemic stroke, and by extension, time to therapy in treated patients and time to transfer from the department for all patients. A secondary objective is to determine if using CTP/CTA-inclusive hyperacute stroke guidelines improves safety by decreasing symptomatic intracerebral hemorrhage and mortality in patients who receive rt-PA.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency Signs and symptoms of acute ischemic stroke: impairment of language, motor function, cognition and/or gaze, vision or neglect.
* Patients with an NIH Stroke Scale score > 4

Exclusion Criteria:

* Age less than 19
* Patient symptomatic for greater than five hours. Intravenous thrombolytic therapy must be instituted within three hours of symptom onset in order to minimize the risk of Intracerebral or symptomatic hemorrhage; other interventions such as intra-arterial thrombolytic therapy and clot retrieval allow for a six-hour window. One hour is an achievable time for arrival to institution of therapy, therefore a five-hour limit on enrollment allows the greatest number of patients the possibility of therapy.
* Inability to verify a clear onset of symptoms. As noted, time elapsed since the patient's last known baseline state is correlated to Intracerebral and symptomatic hemorrhage, and therapy is approved only for patients with a clear time of onset.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Emergency Department with acute stroke
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States